CLINICAL TRIAL: NCT00613548
Title: Moderate Mitral Regurgitation in CABG Patients
Acronym: MoMIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Per Wierup MD, PhD, Assoc Prof, Dep of Cardiothoracic Surgery, Aarhus University Hospital, Skejby, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MoMIC; 20040224
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2008-11-11 (Estimated); Status verified 2008-11

CONDITIONS: Moderate Mitral Regurgitation
Keywords: Moderate; Mitral; Regurgitation; CABG
MeSH Terms: conditions — Lymphoma, Follicular; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): CABG Alone
  Interventions: Procedure: CABG alone
- 2 (Active Comparator): CABG + Mitral repair
  Interventions: Procedure: CABG + Mitral repair

INTERVENTIONS:
Procedure: CABG alone — CABG alone
  Arms: 1
Procedure: CABG + Mitral repair — CABG + Mitral repair
  Arms: 2

SUMMARY:
Background:

The presence of a mild to moderate ischemic mitral regurgitation (IMR) results in a significantly reduced long-term survival and increased hospitalizations for heart-failure. The benefit of adding mitral valve surgery to coronary artery by-pass surgery (CABG) is well documented in the combination of coronary artery disease and severe MR. On the other hand, it is clinical practice to refrain from repairing the mitral valve in those CABG cases where the IMR is mild to moderate. However, there are no conclusive data available to support this principle. The existing studies are small, retrospective, and the results contradictive. The need for a prospective randomized trial has frequently been proposed and discussed, however, to the best of our knowledge, such a study has not yet commenced.

Study design:

The Moderate Mitral Regurgitation In Patients Undergoing CABG (MoMIC) Trial is the first international multi-center, large-scale study to clarify whether moderate IMR in CABG patients should be corrected. A total of 550 CABG patients with moderate IMR are to be randomized to either CABG alone or CABG plus mitral valve correction.

Implication:

If correction of moderate MR in CABG patients is the superior strategy, this should be offered to all patients in this entity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic heart disease, who fulfil the indications for CABG, and who also have a moderate ischemic MR. Ischemic MR is defined as mitral regurgitation due to coronary artery disease and not fortuitously associated with it. It is caused either by a mitral annular dilatation (Carpentier type I), or a restrictive motion of the posterior mitral leaflet (Carpentier type IIIb), or a combination of these. The mitral leaflets should be slender and without signs of intrinsic organic disease. The mitral annulus should be with no significant calcification that can be held responsible for valve insufficiency. The severity of mitral regurgitation is quantified by means of echoardiography using the Proximal Isovelocity Surface Area (PISA)-method. Moderate MR is defined as a calculated ERO of 15-30 mm2 at rest . Hence, patients referred for CABG and showing signs of mitral regurgitation on auscultation, by echocardiography, or by ventriculography will further be evaluated by a thorough echocardiography (Transthoracic (TTE) in ambiguous cases supplemented by transesophageal echocardiography (TEE) before surgery, in order to determine whether the patient fulfil the inclusion criteria. In addition, ejection fraction (visually estimated), left atrial dimension, mitral annular and tricuspid annular size, as well as estimates of pulmonary hypertension will be recorded.
* Age ≥ 18 yrs.
* The inclusion is independent of the left ventricular function.
* The inclusion is independent of the left atrial size.
* It is mandatory that the patient is able to fully understand the written information, the purpose of the study, and able to give an informed consent.

Exclusion Criteria:

* Patients with previous cardiac surgery.
* Emergency surgery.
* Malignant disease with an expected survival of less than 5 years.
* ST-elevation myocardial infarction within 16 days.
* Significant aortic valve disease necessitating aortic valve replacement
* Calcification of the ascending aorta.
* Significant mitral annular calcification.
* Type II MR (ruptured papillary muscle, or infracted elongated papillary muscle with prolapse)
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Death or rehospitalization for heart failure | 5 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Per N Wierup, MD, PhD, Principal Investigator — Dep. of Cardiothoracic Surgery, Aarhus University Hospital, Skejby, Denmark
Locations (1):
- Dep. of Cardiothoracic Surgery, Aarhus University Hospital, Skejby,, Aarhus, Denmark